CLINICAL TRIAL: NCT00864799
Title: Comparison of 3 Regimens Using Mifepristone and Misoprostol for Second Trimester Pregnancy Interruption.
Brief Title: Techniques to Improve Efficacy of Second Trimester Medical Termination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jan Dickinson, Professor Maternal Fetal Medicine, King Edward Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1624/EW
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Pregnancy
Keywords: Abortion; Misoprostol; Mifepristone; Pregnancy; Fetus
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vaginal misoprostol (Active Comparator): Women allocated to the vaginal misoprostol management protocol will receive a loading dose of 800 mcg misoprostol vaginally followed in 4 hours by 400 mcg vaginal misoprostol, the latter repeated every 4 hours for a maximum of 4 doses.
  If abortion does not occur within 24 hours of commencement of this regimen, the sequence will be repeated.
  If delivery is not accomplished within 48 hours of prostaglandin commencement, a transcervical Foley catheter will be inserted and a solution of prostaglandin F2 alpha infused 2-hourly until delivery occurs.
  Interventions: Drug: Misoprostol
- Oral misoprostol (Active Comparator): Women allocated to the standard management protocol will receive a loading dose of 800 mcg misoprostol vaginally followed in 3 hours by 400 mcg misoprostol orally, the latter repeated every 3-hours to a maximum of 4 oral doses.
  If abortion does not occur within 24 hours of commencement of this regimen, the sequence will be repeated.
  If delivery is not accomplished within 48 hours of prostaglandin commencement, a transcervical Foley catheter will be inserted and a solution of prostaglandin F2 alpha infused 2-hourly until delivery occurs.
  Interventions: Drug: Misoprostol
- Sublingual misoprostol (Active Comparator): Women allocated to the sublingual misoprostol protocol will receive a loading dose of 800 mcg misoprostol vaginally followed in 3 hours by 400 mcg sublingual misoprostol, the latter repeated every 3 hours for a maximum of 4 doses.
  If abortion does not occur within 24 hours of commencement of this regimen, the sequence will be repeated.
  If delivery is not accomplished within 48 hours of prostaglandin commencement, a transcervical Foley catheter will be inserted and a solution of prostaglandin F2 alpha infused 2-hourly until delivery occurs.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Comparison of 3 routes of administration of misoprostol for termination of pregnancy 14-24 weeks

SUMMARY:
Interruption of a pregnancy after 14 weeks gestation may be required when the fetus is dead, severely malformed or in cases of maternal illness. This process is usually conducted medically in Australia, using the synthetic prostaglandin E1 analogue misoprostol. This prostaglandin, although not licensed for use in pregnancy termination, is now a common abortifacient with a large accumulated experience both within Australia and internationally. Since 1996, misoprostol has been used at King Edward Memorial Hospital as the principal agent for second trimester pregnancy termination.

Misoprostol may be administered vaginally, orally, sublingually or buccally in the process of pregnancy termination. Each route of administration has its own advantages and disadvantages. The most appropriate route of administration, with the shortest duration of abortion and lowest side-effect profile has not been determined for all circumstances.

The combination of mifepristone and misoprostol is an established and effective method for second trimester pregnancy termination. Prior studies have demonstrated a significant reduction in the duration of abortion with misoprostol when mifepristone priming is used. In November 2007, the TGA (Therapeutic Goods Administration) approved an application by the Principal Investigator of this planned study for Authorised Prescriber status for use of the antiprogesterone agent mifepristone. Since January 2008 the combination of mifepristone and misoprostol has been used at KEMH for first and second trimester pregnancy termination of pregnancy, predominantly for circumstances of severe fetal abnormality.

There is however limited data on the impact of gestation on the duration of second trimester termination. Almost all published studies to date have recruited women in the early second trimester (typically with a median of 16 weeks gestation). However, most terminations of pregnancy for fetal abnormality (the most frequent reason for pregnancy interruption of a live fetus at KEMH) occur at 18-24 weeks gestation. The investigators' experience indicates a significant impact of increasing gestation with prolongation of the duration of pregnancy termination. In this study the investigators aim to evaluate three misoprostol regimens for second trimester pregnancy termination following mifepristone priming with the primary intention to develop a protocol which results in a delivery rate within 24 hours for 95% of women at gestations <24 weeks.

Secondary aims of this study will be to assess the incidence of maternal side-effects for each of the three regimens, the placental retention rates and the need for curettage for retained placental tissue. As the investigators will be using 3 different methods of misoprostol administration, the investigators will also review women's satisfaction with the three regimens for pregnancy termination.

DETAILED DESCRIPTION:
Aims:

1. To compare the efficacy of the vaginal and sublingual administration of the synthetic prostaglandin misoprostol with the currently used vaginal administration route in second trimester pregnancy termination.
2. To compare the impact of gestation of the duration of abortion within these three misoprostol regimens.
3. To compare the incidence of maternal side-effects between the three routes of prostaglandin administration.
4. To compare the incidence of placental retention and need for curettage between the three groups

ELIGIBILITY:
Inclusion Criteria:

* 14-24 weeks pregnant
* planned medical termination
* able to speak and understand English
* no contraindication to prostaglandins

Exclusion Criteria:

* gestation < 13 weeks
* allergy/contraindication to misoprostol
* allergy/contraindication to mifepristone
* fetal demise

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 302 (Actual)
Dates: Start 2009-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of the vaginal and sublingual administration of the synthetic prostaglandin misoprostol with the currently used oral administration route in second trimester pregnancy termination. | Induction to delivery interval

SECONDARY OUTCOMES:
To compare the incidence of maternal side-effects between the three routes of prostaglandin administration. | Admission to hospital discharge
To compare the incidence of placental retention and need for curettage between the three groups | Delivery of fetus to delivery of placenta interval
To compare the impact of gestation of the duration of abortion within these three misoprostol regimens. | Interval from commencement of prostaglandin to delivery of fetus

CONTACTS AND LOCATIONS:
Overall Officials: Jan E Dickinson, MD, Principal Investigator — The University of Western Australia
Locations (1):
- King Edward Memorial Hospital, Perth, Western Australia, Australia

REFERENCES:
- [Derived] Dickinson JE, Jennings BG, Doherty DA. Mifepristone and oral, vaginal, or sublingual misoprostol for second-trimester abortion: a randomized controlled trial. Obstet Gynecol. 2014 Jun;123(6):1162-1168. doi: 10.1097/AOG.0000000000000290. PMID 24807339